CLINICAL TRIAL: NCT00883324
Title: A Phase IIIB Comparison of Fetal Fibronectin (fFN) Specimen Collection Methodologies: With Speculum Versus Without Speculum
Brief Title: Comparison of Fetal Fibronectin (fFN) Specimen Collection Methodologies: With Speculum Versus Without Speculum
Acronym: SpecOp
Status: Completed | Type: Observational
Sponsor: Hologic, Inc. (Industry)
Responsible Party: Arthur Friedman, Senior Vice President of Quality, Regulatory and Clinical, Hologic
Other Study IDs: D0108001
Record Dates: First submitted 2009-04-10; First posted 2009-04-17 (Estimated); Last update posted 2011-06-20 (Estimated); Status verified 2011-06

CONDITIONS: Preterm Delivery
Keywords: fFN; fetal fibronectin; non-speculum; risk of preterm delivery
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: fetal fibronectin specimens collected with a speculum
- 2: fetal fibronectin specimens collected without a speculum

SUMMARY:
Observational study to determine whether the proposed method of fFN specimen collection without a speculum is substantially equivalent to the approved method with a speculum examination when obtained at the gestational age of ≥ 24 weeks and ≤ 34, 6 days in symptomatic women and at the gestational age of ≥ 22 weeks, 0 days and ≤ 30, 6 days in asymptomatic women. A finding of substantial equivalency would support a modification to the labeling to allow the collection of specimens for fFN determination with or without a speculum examination.

DETAILED DESCRIPTION:
The study population will include pregnant women who may be at risk for preterm delivery and require the fFN test, as determined by their doctor to aid in patient management. The subjects may or may not present with symptoms related to preterm labor and must satisfy the device's approved labeling and the eligibility criteria.

For pregnant women with signs of labor, the Fetal Fibronectin (fFN) test is approved for use as an aid to assess the risk of preterm delivery in ≤ 7 or ≤ 14 days from cervicovaginal sample collection that have intact amniotic membranes and minimal cervical dilation (< 3 cm) and are sampled between 24 weeks, 0 days and 34 weeks, 6 days. It is also approved for use with additional clinical information in asymptomatic women with singleton pregnancies when a sample is obtained during a routine prenatal visit between 22 weeks, 0 days and 30 weeks, 6 days of gestation.

The fFN test is run on The Rapid fFN for the TLiIQ® System and a positive fFN result occurs with concentrations ≥50ng/mL and a negative fFN test with concentrations <50ng/mL.

The current FDA-approved labeling for the collection of the fFN specimen requires a speculum examination; however, the collection of the fFN specimen is often needed when the women first arrives at the hospital labor and delivery unit, where nurses often are not trained or credentialed to perform speculum examinations and a physician may not be readily available to perform the collection. Therefore, there is an unmet need for a simpler collection method.

The test article in this study is the collection of cervicovaginal samples for fFN determination using a standardized collection method without a speculum. The control article in this study is the collection of a cervicovaginal sample for fFN determination using the approved collection method requiring a speculum examination. Both the test and control fFN specimen samples will be collected and evaluated using the approved Rapid fFN for the TLiIQ® System.

The primary objective of this study is to determine whether the proposed method of fFN specimen collection without a speculum is substantially equivalent to the approved method with a speculum examination when obtained at the gestational age of ≥ 24 weeks and ≤ 34, 6 days in symptomatic women and at the gestational age of ≥ 22 weeks, 0 days and ≤ 30, 6 days in asymptomatic women. A finding of substantial equivalency would support a modification to the labeling to allow the collection of specimens for fFN determination with or without a speculum examination.

Hypothesis: The method of fFN specimen collection without a speculum is not inferior to collection with a speculum within a 5% margin of non-inferiority.

ELIGIBILITY:
Inclusion Criteria:

* Maternal age > 18 years.
* Subject has signed and dated an Institutional Review Board (IRB) or Research Ethics Board (REB) approved consent form to participate in the study.
* Specimen Collection Kit and the Rapid fFN for the TLiIQ® System are currently utilized as standard of care (SOC).
* Gestational age of ≥ 24 weeks, 0 days and ≤ 34 weeks, 6 days for symptomatic subjects. (As defined by ACOG.)
* Gestational age of ≥ 22 weeks, 0 days and ≤ 30 weeks, 6 days for asymptomatic subjects with singleton pregnancies. (As defined by ACOG.)
* Intact amniotic membranes.

Exclusion Criteria:

* Placenta previa or abruptio placenta.
* Cervical cerclage.
* Digital examination, vaginal intercourse, or transvaginal ultrasound within 24 hours prior to the fFN sample collection.
* Moderate or gross vaginal bleeding at the time of fFN sample collection. Cervical dilatation ≥ 3 centimeters.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Labor and delivery triage, prenatal clinic
Sampling Method: Non-Probability Sample
Enrollment: 329 (Estimated)
Dates: Start 2009-03

CONTACTS AND LOCATIONS:
Overall Officials: James D. Byrne, M.D., Principal Investigator — Santa Clara Valley Medical Health & Hospital System; Michael Paidas, M.D., Principal Investigator — Yale University; Larry Matsumoto, M.D., Principal Investigator — Northside Hospital Center for Perinatal Medicine; Janice Whitty, MD, Principal Investigator — Meharry Medical College; John Allbert, MD, Principal Investigator — Presbyterian Hospital; Annette E. Bombrys, DO, Principal Investigator — Kettering Health Network
Locations (5):
- United States (5):
  - Santa Clara Valley Medical Health & Hospital System, San Jose, California
  - Yale University Medical Center, New Haven, Connecticut
  - Northside Hospital, Atlanta, Georgia
  - Presbyterian Hospital, Charlotte, North Carolina
  - Kettering Health Network of Kettering Medical Center, Kettering, Ohio